CLINICAL TRIAL: NCT06965218
Title: Relation Between Aortic Valve Sclerosis and Severity of Coronary Heart Disease Assessed by Syntax Score in Sohag University Hospital
Brief Title: Relation Between Aortic Sclerosis &Severity of Coronary Heart Disease.
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Aly Mohamed, cardiologist, Sohag University
Other Study IDs: Soh-Med-25-4___1MD
Record Dates: First submitted 2025-04-24; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Aortic Valve Sclerosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Trans thoracic echo doppler — Aortic valve sclerosis severity study be transthoracic echo doppler

SUMMARY:
the goal of the study to identify the relation between aortic valve sclerosis and severity of coronary heart disease by performing transthoracic echo Doppler study for severity of aortic valve sclerosis in patient will undergo coronary angiography with calculation of syntax score as a tool for severity of coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Aortic sclerosis diagnosed by trans thoracic echo doppler

Exclusion Criteria:

* patients who known to be Rumatic heart disease or congenital aortic valve disease.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 100a patients from both sex who are diagnosed to be aortic valve sclerosis and will undergo coronary angiography in Sohag university hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
relation between Aortic valve sclerosis and severity of coronary heart disease | 6 months
  significant relation between severity of aortic valve sclerosis assessed by trans thoracic echo doppler quantified by Chandra et al on a scale of 0 to 3.
  0 (no involvement).
  1. mild (minor involvement of one leaflet)
  2. moderate (minor involvement of two leaflets or extensive involvement of one leaflet.
  3. severe (extensive involvement of two leaflets or involvement of all three leaflets).
  And severity of coronary heart disease in patients already underwent or planned to perform coronary angiography quantified by syntax score considering score above 20 as severe coronary heart disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt